CLINICAL TRIAL: NCT06509386
Title: Randomized Vignette Experiment on the Effects of Portrayals of Successful Treatment and Role Fulfillment on Mental Illness Stigma
Brief Title: Effects of Portrayals of Successful Treatment and Role Fulfillment on Mental Illness Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000034605_b
Record Dates: First submitted 2024-06-07; First posted 2024-07-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Mental Illness
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Major Depressive Disorder without treatment or role fulfillment (Experimental)
  Interventions: Other: Major Depressive Disorder without treatment or role fulfillment
- Major Depressive Disorder with treatment but no role fulfillment (Experimental)
  Interventions: Other: Major Depressive Disorder with treatment but no role fulfillment
- Major Depressive Disorder without treatment but with role fulfillment (Experimental)
  Interventions: Other: Major Depressive Disorder without treatment but with role fulfillment
- Major Depressive Disorder with treatment and role fulfillment (Experimental)
  Interventions: Other: Major Depressive Disorder with treatment and role fulfillment
- Schizophrenia without treatment or role fulfillment (Experimental)
  Interventions: Other: Schizophrenia without treatment or role fulfillment
- Schizophrenia with treatment but no role fulfillment (Experimental)
  Interventions: Other: Schizophrenia with treatment but no role fulfillment
- Schizophrenia without treatment but with role fulfillment (Experimental)
  Interventions: Other: Schizophrenia without treatment but with role fulfillment
- Schizophrenia with treatment and role fulfillment (Experimental)
  Interventions: Other: Schizophrenia with treatment and role fulfillment

INTERVENTIONS:
Other: Major Depressive Disorder without treatment or role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Major Depressive Disorder without treatment or role fulfillment
Other: Major Depressive Disorder with treatment but no role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Major Depressive Disorder with treatment but no role fulfillment
Other: Major Depressive Disorder without treatment but with role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Major Depressive Disorder without treatment but with role fulfillment
Other: Major Depressive Disorder with treatment and role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Major Depressive Disorder with treatment and role fulfillment
Other: Schizophrenia without treatment or role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Schizophrenia without treatment or role fulfillment
Other: Schizophrenia with treatment but no role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Schizophrenia with treatment but no role fulfillment
Other: Schizophrenia without treatment but with role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Schizophrenia without treatment but with role fulfillment
Other: Schizophrenia with treatment and role fulfillment — Read vignette describing the condition and ask stigma questions.
  Arms: Schizophrenia with treatment and role fulfillment

SUMMARY:
This study aims to measure levels of mental illness stigma based on successful treatment and societal role fulfillment of the individual portrayed with mental illness.

DETAILED DESCRIPTION:
This study aims to measure levels of mental illness stigma based on successful treatment and societal role fulfillment of the individual portrayed with mental illness. This study utilizes eight vignettes portraying two different mental illnesses (depression and schizophrenia), with one vignette giving no details about role fulfillment or treatment, another giving no details about role fulfillment but successful treatment, another giving details on role fulfillment but no treatment, and last giving details on both role fulfillment and successful treatment.

ELIGIBILITY:
Inclusion Criteria:

* All adults who consider Buyende District their primary residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age
* Persons who do not consider Buyende District their primary place of residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Personal Acceptance Scale (PAS) | One year. For each interview, approximately 60 minutes.
  The PAS is a questionnaire targeted to public stigma, the "negative attitudes, beliefs, and behaviors held within a community" against individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. There were ten questions, therefore it generated a score between zero and ten. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.
Broad Acceptance Scale (BAS) | One year. For each interview, approximately 60 minutes.
  The BAS is a questionnaire targeted to distal public stigma. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. There were ten questions, therefore it generated a score between zero and ten. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.
Attributed Stigma Scale | One year. For each interview, approximately 60 minutes.
  Attributed stigma scale will be a modification of the PAS to gather understanding of what participants believe the attitudes of others in their community are. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. There were ten questions, therefore it generated a score between zero and ten. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jae Lee, MD, Principal Investigator — Yale University
Locations (1):
- Empowerment to Heal - Uganda, Iganga, Uganda

IPD SHARING:
Plan to Share IPD: No